CLINICAL TRIAL: NCT03372889
Title: On-Q Catheter Caregiver Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-0638
Record Dates: First submitted 2017-12-01; First posted 2017-12-14 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Anterior Cruciate Ligament Injury; Pain; Catheter (Other); Satisfaction, Personal
Keywords: Anterior Cruciate Ligament; On-Q Catheter; nerve block; ACL reconstruction; patient education materials
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Subjects are randomized into one of the following two groups:
  Group 1: Print based PEM Group 2: Media based PEM All study outcomes are compared between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient educaiton materials Print based (Active Comparator): Patients are randomly assigned to view print based educational material.
  Interventions: Behavioral: Patient educaiton materials - Print based
- Patient educaiton materials Media Based (Active Comparator): Patients are randomly assigned to view media based educational material.
  Interventions: Behavioral: Patient educaiton materials - Media based

INTERVENTIONS:
Behavioral: Patient educaiton materials - Print based — Print (paper) based materials
  Other Names: Print based
  Arms: Patient educaiton materials Print based
Behavioral: Patient educaiton materials - Media based — Media (electronic) based materials
  Other Names: Media based
  Arms: Patient educaiton materials Media Based

SUMMARY:
The present study aims to compare caregiver satisfaction and efficacy between two modes of patient education materials (PEMs): media based and print based. The caregivers of patient's who undergo ACL (anterior cruciate ligament) reconstruction surgery and receive an On-Q Catheter pain block receive both a hand-out (print based PEM) and watch a short video (media-based PEM) describing how to care for their child's On-Q Catheter at home. Upon enrollment into the study, caregivers are randomly assigned to either first view the hand-out or the video, then complete a 10 questions standardized assessment of information that was presented in the PEMs. Caregivers are called the next day to assess caregiver satisfaction with the PEMs, which mode of PEM was more helpful to them, and how comfortable they felt managing their child's pain pump at home.

DETAILED DESCRIPTION:
The present study aims to compare the efficacy and caregiver satisfaction between two modes of patient education materials (PEMs): media based and print based. The PEMs are designed to education caregivers on how to manage their child's On-Q catheter pain block at home. After caregivers have enrolled in the study and have been randomized to an education group, study interventions take place in the private family waiting room. Immediately after viewing their assigned PEM, the caregiver completes a 10 question standardized assessment, formatted as a multiple-choice quiz, of their understanding and knowledge of the information conveyed in both modes of PEM. The following day, caregivers are contacted by phone call to answer a number of questions to assess their satisfaction with the PEMs they received, the mode of PEM they preferred, and how comfortable they felt managing their child's pain pump at home.

All information is stored in a secure database (REDCap).

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of patients undergoing ACL repair/reconstruction. These caregivers are registered in the Children's Hospital of Colorado medical record.

Exclusion Criteria:

* Illiterate or blind individuals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with Patient Education Materials (PEM). | Twenty-four to 48 hours post-operatively
  Determine whether one of these forms, print-based PEMs or media-based PEMs, results in greater patient satisfaction versus the other.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa N Mandler, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided